CLINICAL TRIAL: NCT01268969
Title: A Prospective Randomized Trial-comparing Excision and Limberg Flap Closure Versus Karydakis Flap Reconstruction for Treatment of Sacrococcygeal Pilonidal Disease
Brief Title: Comparison Between Two Different Technique in Treatment of Chronic Pilonidal Disease
Acronym: PND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: WALEED ASKAR, mansoura university hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMRO-1234
Record Dates: First submitted 2010-12-29; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2008-02

CONDITIONS: Pilonidal Disease
Keywords: pilonidal disease PND

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- excision and krydakis reconstruction (Active Comparator): The technique consisted of a vertical eccentric elliptical incision carried down to the post sacral fascia, complete removal of unhealthy tissue with the normal tissue around the cyst and sinus tracts, mobilization of the medial wound edge by undercutting the adipose tissue at a depth of 1 cm, the advancement of the flap across the midline to the post sacral fascia and suturing of its edge to the lateral one
  Interventions: Procedure: KARYDAKIS GROUP
- surgical excision and limberg closure (Active Comparator): The area to be excised was mapped on the skin in a rhomboid form . The skin incision was deepened to the presacral fascia centrally and to the gluteal fascia laterally. After removing the specimen, the Limberg fasciocutaneous flap was prepared by extending the incision down to and through the right gluteus maximus fascia . The fasciocutaneous flap was transposed medially so that the defect would be covered without any tension.
  Interventions: Procedure: Lamberg flap technique

INTERVENTIONS:
Procedure: KARYDAKIS GROUP — The technique consisted of a vertical eccentric elliptical incision carried down to the post sacral fascia, complete removal of unhealthy tissue with the normal tissue around the cyst and sinus tracts, mobilization of the medial wound edge by undercutting the adipose tissue at a depth of 1 cm, the advancement of the flap across the midline to the post sacral fascia and suturing of its edge to the lateral one
  Other Names: GROUP 1
  Arms: excision and krydakis reconstruction
Procedure: Lamberg flap technique — The area to be excised was mapped on the skin in a rhomboid form . The skin incision was deepened to the presacral fascia centrally and to the gluteal fascia laterally. After removing the specimen, the Limberg fasciocutaneous flap was prepared by extending the incision down to and through the right gluteus maximus fascia
  Other Names: group 2
  Arms: surgical excision and limberg closure

SUMMARY:
Comparison between limberg flap and Karydakis flap for treatment of pilonidal disease.

DETAILED DESCRIPTION:
The authors prospectively studied patients with sacrococcygeal pilonidal disease (SPD) at Mansoura University Hospital, Mansoura, Egypt, .Patients were randomly assigned to undergo either Limberg rhomboid flap or Karydakis flap reconstruction . The follow-up period ranged from 8 months to two years, with the mean follow-up period about 18 months. Surgical findings, complications, recurrence rate and degree of patient satisfaction were compared. This a randomized controlled study to evaluate both rhomboid excision and limberg flap closure versus Karydakis flap for treatment of chronic pilonidal disease.

Karydakis flap reconstruction was performed in conformity with the original procedure described by Karydakis. The technique consisted of a vertical eccentric elliptical incision carried down to the post sacral fascia, complete removal of unhealthy tissue with the normal tissue around the cyst and sinus tracts, mobilization of the medial wound edge by undercutting the adipose tissue at a depth of 1 cm, the advancement of the flap across the midline to the post sacral fascia and suturing of its edge to the lateral one.

Lamberg flap technique: the area to be excised was mapped on the skin in a rhomboid form . The skin incision was deepened to the presacral fascia centrally and to the gluteal fascia laterally. After removing the specimen, the Limberg fasciocutaneous flap was prepared by extending the incision down to and through the right gluteus maximus fascia (Fig3a). The size of the prepared flap was equal to that of the rhomboid area. Meticulous hemostasis was accomplished by electrocauterization. The fasciocutaneous flap was transposed medially so that the defect would be covered without any tension. Sutures were placed between gluteus fascia of the flap and presacral fascia with 2/0 polyglactin to prevent dead space

ELIGIBILITY:
Inclusion Criteria:

* PATINTS WITH PILONIDAL SINUS

Exclusion Criteria:

* PILONIDAL ABSCESS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
EARLY COMPLICATIONS , HEALING , EARLY RETURN TO WORK | 2 years
  efficacy of the procedures , short and long term patients satisfactions

CONTACTS AND LOCATIONS:
Overall Officials: waleed askar, M.D, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Result] Topgul K, Ozdemir E, Kilic K, Gokbayir H, Ferahkose Z. Long-term results of limberg flap procedure for treatment of pilonidal sinus: a report of 200 cases. Dis Colon Rectum. 2003 Nov;46(11):1545-8. doi: 10.1007/s10350-004-6811-y. PMID 14605577
- [Result] Fuzun M, Bakir H, Soylu M, Tansug T, Kaymak E, Harmancioglu O. Which technique for treatment of pilonidal sinus--open or closed? Dis Colon Rectum. 1994 Nov;37(11):1148-50. doi: 10.1007/BF02049819. PMID 7956585
- [Result] el-Khadrawy O, Hashish M, Ismail K, Shalaby H. Outcome of the rhomboid flap for recurrent pilonidal disease. World J Surg. 2009 May;33(5):1064-8. doi: 10.1007/s00268-009-9920-x. PMID 19198934
- [Result] Mahdy T. Surgical treatment of the pilonidal disease: primary closure or flap reconstruction after excision. Dis Colon Rectum. 2008 Dec;51(12):1816-22. doi: 10.1007/s10350-008-9436-8. Epub 2008 Oct 21. PMID 18937009
- See also: Mansoura university — http://www.mans.eun.eg